CLINICAL TRIAL: NCT00655811
Title: Ethnic Differences in Response to Topical Capsaicin: A Psychophysical Study on Healthy Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 00003739
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Results first posted 2017-08-14 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Healthy
Keywords: Healthy volunteers
MeSH Terms: interventions — Capsaicin; cetyl alcohol, propylene glycol, sodium lauryl sulfate non-lipid cleansing lotion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capsaicin (Active Comparator): Capsaicin 0.1% cream application to the volar side of forearm.
  Interventions: Drug: Capsaicin
- Placebo moisturizing cream (Placebo Comparator): Placebo moisturizing cream with no active ingredient (Cetaphil; Galderma Laboratories LP, Fort Worth, TX, U.S.A.) to the opposite forearm.
  Interventions: Drug: Placebo moisturizing cream

INTERVENTIONS:
Drug: Capsaicin — Topical application, 0.1%, Capzasin HP; Chattem Inc., Chattanooga, TN, U.S.A
  Other Names: Topical capsaicin, 0.1%, Capzasin HP
  Arms: Capsaicin
Drug: Placebo moisturizing cream — Placebo moisturizing cream with no active ingredient (Cetaphil; Galderma Laboratories LP, Fort Worth, TX, U.S.A.)
  Other Names: Cetaphil
  Arms: Placebo moisturizing cream

SUMMARY:
The purpose of this research is to study how people respond differently to capsaicin in different racial groups and the effect it has on your pain levels. Capsaicin is a natural product made from hot chili peppers that is useful for treating the itch symptoms of skin disease.

DETAILED DESCRIPTION:
To comprehensively evaluate the ethnic differences in response to topical capsaicin and its effect on thermal sensory thresholds.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women who are between 18 and 50 years of age.
* Subjects must be in general good health with no skin disease, disease state or physical condition which would impair evaluation of pain perception or which would increase their health risk by study participation as determined by the investigators.
* Women of childbearing potential will be required to have a negative pregnancy test in order to enroll in the study.

Exclusion Criteria:

* Adults over age 50.
* Children less than 18 years of age.
* Unable to complete the required measures.
* Diagnosis of diseases that would affect the measurement of pain perception.
* Currently enrolled in any investigational study in which the subject is receiving any type of drug, biologic, or non-drug therapy and subjects undergoing treatment with another investigational drug or approved therapy for investigational use within 30 days prior to study participation.
* Use of oral analgesic or other medications known to interfere with pain perception in the week prior to the study.
* Use of emollient on the forearms on the day of the study visit.
* Use of medicated topical preparations on the forearms for the week prior to the study.
* Known history of neuropathy causing diseases such as uremia.
* Known history of uncontrolled thyroid disease.
* Known history of diabetes mellitus.
* Allergy to capsaicin.
* Pregnant women.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-02; Primary Completion 2008-08 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gil Yosipovitch, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences Dermatology, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Capsaicin and Placebo: 0.1% Topical Capsaicin cream was applied to one forearm and a placebo moisturizing cream with no active ingredient (Cetaphil; Galderma Laboratories LP, Fort Worth, TX, U.S.A.) was applied to the other forearm.
  A volume of 0·3 mL cream was applied in a thin layer of virtually equal thickness, on a 4 × 4 cm area, around midline. The creams were applied at a 40-min interval in a random order to minimize an order effect. The creams were randomized for right and left arm application.
Period: Overall Study
Arm/Group | Capsaicin and Placebo
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Capsaicin and Placebo: 0.1% Topical Capsaicin cream was appled to one forearm and a placebo moisturizing cream with no active ingredient (Cetaphil; Galderma Laboratories LP, Fort Worth, TX, U.S.A.) was applied to the other forearm.
  A volume of 0·3 mL cream was applied in a thin layer of virtually equal thickness, on a 4 × 4 cm area, around midline. The creams were applied at a 40-min interval in a random order to minimize an order effect. The creams were randomized for right and left arm application.
Arm/Group | Capsaicin and Placebo
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African Americans | 10
  Caucasians | 10
  East Asians | 10
  Hispanic | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Ethnic Differences in Burning Pain Induced by Topical Capsaicin
Description: The primary endpoint is to test the burning pain effect of topical capsaicin by using an continuous visual analog scale (CoVAS) intensity scale as an outcome measure. Participants will rate burning pain intensity after topical capsaicin application. The burning or pain sensation intensity was recorded continuously on a 100-mm COVAS (0, no sensation to 100, maximum, strongest imaginable pain sensation). The subjects were also asked to indicate whether they experienced any nonpainful sensation.
Time Frame: 1 day
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- African Americans; Caucasians; East Asians; Hispanics: 0.1% Topical Capsaicin cream was applied to one forearm and a placebo moisturizing cream with no active ingredient (Cetaphil; Galderma Laboratories LP, Fort Worth, TX, U.S.A.) was applied to the other forearm.
  A volume of 0·3 mL cream was applied in a thin layer of virtually equal thickness, on a 4 × 4 cm area, around midline. The creams were applied at a 40-min interval in a random order to minimize an order effect. The creams were randomized for right and left arm application.
Arm/Group | African Americans | Caucasians | East Asians | Hispanics
Number analyzed (Participants) | 10 | 10 | 10 | 10
units on a scale
  Capsaicin | 0.81 (0.68) | 4.07 (1.61) | 17.05 (5.80) | 13.3 (4.67)
  Placebo | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Statistical Analysis 1: Comparison: African Americans vs Caucasians vs East Asians vs Hispanics; One-way anova was used to compare the mean COVAS values between groups; Test type: Superiority; p < 0.05, ANOVA
Statistical Analysis 2: Comparison: African Americans vs Caucasians; Test type: Superiority; p = 0.550, t-test, 2 sided
Statistical Analysis 3: Comparison: African Americans vs East Asians; Test type: Superiority; p = 0.005, t-test, 2 sided
Statistical Analysis 4: Comparison: African Americans vs Hispanics; Test type: Superiority; p = 0.027, t-test, 2 sided

2. Secondary Outcome: Ethnic Differences on the Effects of Topical Capsaicin on Thermal Sensory Thermal Thresholds
Description: A secondary endpoint is to see if topical capsaicin has an effect on warm and heat pain thresholds. Quantitative thermosensory testing was carried out using the Medoc TSA 2001 (Medoc Ltd). The probe baseline temperature was 32 °C and the contact area was 12 cm2. The probe warmed the skin surface at a linear rate of 0·4 °C per second, up to a cut-off of 50 °C. Thermal thresholds were measured in the following order: warmth sensation threshold was measured followed by heat pain detection threshold; each of them was determined four times by the ascending method of limits.
Time Frame: 1 day
Measure: Mean (Standard Error); unit: Change in degrees Celsius
Arm/Group | African Americans | Caucasians | East Asians | Hispanics
Number analyzed (Participants) | 10 | 10 | 10 | 10
Change in degrees Celsius
  Heat pain detection threshold change | -2.11 (1.12) | -6.10 (1.36) | -5.01 (1.09) | -7.24 (0.57)
  Warmth sensation threshold change | 2.36 (0.93) | -0.68 (0.68) | 0.56 (.059) | -3.15 (0.93)
Statistical Analysis 1: Comparison: African Americans vs Caucasians; Test type: Superiority; p = 0.012, t-test, 2 sided
Statistical Analysis 2: Comparison: African Americans vs East Asians; Test type: Superiority; p = 0.06, t-test, 2 sided
Statistical Analysis 3: Comparison: African Americans vs Hispanics; Test type: Superiority; p = 0.002, t-test, 2 sided

3. Secondary Outcome: The Difference in Burning/Pain Sensation Ratings Between the Capsaicin or Placebo Application.
Description: This secondary outcome is to see if subjects rated burning/pain differently between the topical capsaicin or placebo application. Participants will rate burning/pain intensity after topical capsaicin and placebo application. The burning/pain sensation intensity was recorded continuously on a 100-mm COVAS (0, no sensation to 100, maximum, strongest imaginable burning/pain sensation). The subjects were also asked to indicate whether they experienced any non-burning/-painful sensation.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Capsaicin: 0.1% Topical Capsaicin cream was applied to one forearm.
  A volume of 0·3 mL cream was applied in a thin layer of virtually equal thickness, on a 4 × 4 cm area, around midline. The creams were applied at a 40-min interval in a random order to minimize an order effect. The creams were randomized for right and left arm application.
- Placebo: A placebo moisturizing cream with no active ingredient (Cetaphil; Galderma Laboratories LP, Fort Worth, TX, U.S.A.) was applied to the other forearm.
  A volume of 0·3 mL cream was applied in a thin layer of virtually equal thickness, on a 4 × 4 cm area, around midline. The creams were applied at a 40-min interval in a random order to minimize an order effect. The creams were randomized for right and left arm application.
Arm/Group | Capsaicin | Placebo
Number analyzed (Participants) | 40 | 40
units on a scale | 8.81 (7.63) | 0 (0)
Statistical Analysis 1: Comparison: Capsaicin vs Placebo; Test type: Superiority; p = 0.06, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Capsaicin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes